CLINICAL TRIAL: NCT06747039
Title: ObServational StUdy of CaNnabis ExtRact in FIbromyalgia SyndromE
Brief Title: Cannabis Extract in Fibromyalgia Syndrome - the SUNRISE Study
Acronym: SUNRISE
Status: Recruiting | Type: Observational
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Other Study IDs: SUNRISE (L4184)
Record Dates: First submitted 2024-12-18; First posted 2024-12-24 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Fibromyalgia (FM)
Keywords: fibromyalgia; cannabis; pain; fatigue; quality of life; sleep disturbances
MeSH Terms: conditions — Fibromyalgia; Marijuana Abuse; Pain; Fatigue; Parasomnias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with a diagnosis of FM after failure and/or intolerance of first- and second-line treatment: Patients with a diagnosis of FM according to 2016 American College of Rheumatology Criteria, aged 18 years and older, able to fully understand and fill questionnaires and to provide fully informed consent, who failed and/or were intolerant of first- or second-line treatment.

SUMMARY:
The aim of this observational study is to evaluate the effects of cannabis extract Avextra 10/10 solution on pain, fatigue, sleep, and quality of life among patients affected by fibromyalgia (FM) syndrome. The main question it aims to answer is:

Does cannabis extract have a positive effect on pain after 12 weeks in these patients?

Participants diagnosed from FM will be evaluated and will fill survey about their pain, fatigue, sleep, anxiety, depression and quality of life at baseline, 4 weeks, 8 weeks and 12 weeks after the initiation of cannabis extract Avextra 10/10 solution.

DETAILED DESCRIPTION:
Fibromyalgia (FM) is a chronic condition characterized by widespread pain, mechanical hyperalgesia, fatigue, sleep disturbances, psychological and cognitive impairments, mood changes, headaches, migraines, and gastrointestinal symptoms. Despite its recognition as a medical condition with diagnostic criteria and severity scales, its exact causes and effective treatment remain unclear. FM significantly impacts patients' quality of life and poses a societal burden due to high direct and indirect costs.

Cannabis-based treatments have gained attention for FM symptom management. In Italy, therapeutic cannabis has been legal since 2013 and may be prescribed when conventional treatments fail or cause intolerable side effects. Its primary components, tetrahydrocannabinol (THC) and cannabidiol (CBD), interact with cannabinoid receptors to potentially provide pain relief, anti-inflammatory effects, and mood stabilization.

The study aims to evaluate the efficacy of the standardized cannabis extract Avextra 10/10 (10 mg/mL THC and 10 mg/mL CBD) for FM treatment.

Objectives Primary objective: -Assess the extract's impact on pain after 12 weeks.

Secondary objective:

* Evaluate the clinical effect of cannabis extract Avextra 10/10 solution on fatigue, sleep, anxiety and depression after 4, 8 and 12 weeks among patients affected by FM
* Evaluate the clinical effect of cannabis extract Avextra 10/10 solution on pain after 4 and 8 weeks among patients affected by FM.
* Evaluate the effect of cannabis extract Avextra 10/10 solution on the quality of life at 4, 8 and 12 weeks among patients affected by FM.
* Describe any adverse events or the principal reasons of drug discontinuation.

Design and Methods This is a monocentric observational prospective study in which patients with FM who undertake cannabis therapy with cannabis extract Avextra 10/10 solution will consecutively be recruited.

Population: The inclusion criteria are:

* Patients with a diagnosis of FM according to 2016 American College of Rheumatology Criteria [2].
* Patients with FM prescribed cannabis extract Avextra 10/10 solution after failure and/or intolerance of first- or second-line treatment.
* Aged 18 years and older.
* Able to fully understand and fill questionnaires.
* Able to provide informed consent, according to requirements of local IRB/ethics committee.

The exclusion criteria are:

* Known history of pain not due to FM.
* Patients who have not received stable therapy for pain, sleep disorders, or any psychiatric condition for at least 2 weeks.
* Patients who are taking other types of medical cannabis besides Avextra 10/10 solution.
* Concomitant diagnosis of other pathologies that could interfere with clinical judgment.
* Psychiatric diagnosis according to DSM-V-TR

All patients with FM will undergo a standard clinical assessment, at baseline and at the follow-up visits, as part of the routine clinical practice. After the baseline visit, corresponding to the appointment where medical cannabis is prescribed within two weeks before the undertake of cannabis extract, follow-up visits will be scheduled according to routine clinical practice as follow:

* 15 days after the undertake of cannabis extract (T15)
* 30 days after the undertake of cannabis extract (T30)
* 60 days after the undertake of cannabis extract (T60)
* 90 days after the undertake of cannabis extract (T90)
* 6 months after the undertake of cannabis extract. All patients with FM will undergo a standard clinical assessment, at baseline and at the follow-up visits, as part of the routine clinical practice.

Data collected from participants during clinical evaluations at baseline visit will include:

* Demographic data: age, gender, BMI, residence
* Educational qualification
* Occupational status
* Age at menopause (if applicable)
* Current medication
* Comorbidities
* Symptom duration
* Age at FM diagnosis
* Number of sure tender point
* Smoke status
* Physical activity

Data collected from participants during clinical evaluations at follow-up visit will include:

* Number of sure tender point
* Smoke status
* Physical activity
* Efficacy or side effects of cannabis extract
* Discontinuation of cannabis extract

Conclusion The study seeks to establish the feasibility and clinical effects of a standardized cannabis extract for FM, addressing a critical gap in treatment strategies. Further research is needed to validate its efficacy and optimize FM management.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of FM according to 2016 American College of Rheumatology Criteria.
* Patients with FM prescribed cannabis extract Avextra 10/10 solution after failure and/or intolerance of first- or second-line treatment.
* Aged 18 years and older.
* Able to fully understand and fill questionnaires.
* Able to provide informed consent, according to requirements of local IRB/ethics committee.

Exclusion Criteria:

* Known history of pain not due to FM.
* Patients who have not received stable therapy for pain, sleep disorders, or any psychiatric condition for at least 2 weeks.
* Patients who are taking other types of medical cannabis besides Avextra 10/10 solution.
* Concomitant diagnosis of other pathologies that could interfere with clinical judgment.
* Psychiatric diagnosis according to DSM-V-TR
* Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients afferent to IRCCS Ospedale Galeazzi Sant- Ambrogio in Milan (Italy) with FIbromyalgia Syndrome who will start therapy with cannabis extract Avextra 10/10.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Estimated)
Dates: Start 2024-12-05 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Evaluate the clinical effect of cannabis extract Avextra 10/10 solution on pain after 12 weeks among patients affected by FM | 12 weeks
  The primary endpoint is based on a comparative analysis between the Visual Analogic Scale (VAS) score reported before cannabis extract Avextra 10/10 solution and after 12 weeks of therapy. VAS will use a 100 mm pain line where 0 represents "no pain at all" and 100 is "maximum pain ever experienced".

SECONDARY OUTCOMES:
Evaluate the clinical effect of cannabis extract Avextra 10/10 solution on sleep quality among patients affected by FM using Pittsburgh sleep quality index (PSQI) | 4, 8 and 12 weeks
  Pittsburgh sleep quality index (PSQI) consists of 19 self-rated questions and 5 questions rated by a bed partner or roommate (if applicable).
  The self-rated items are organized into seven component scores:
  * Subjective Sleep Quality: Perceived sleep quality overall.
  * Sleep Latency: Time taken to fall asleep.
  * Sleep Duration: Total hours of actual sleep per night.
  * Habitual Sleep Efficiency: Ratio of actual sleep to time spent in bed.
  * Sleep Disturbances: Frequency of problems such as waking up during the night.
  * Use of Sleep Medication: Frequency of use of sleeping pills or aids.
  * Daytime Dysfunction: Impact of poor sleep on daily activities, such as feeling tired or having difficulty concentrating.
  Each component is scored on a scale of 0 to 3, with higher scores indicating greater difficulty or poorer quality in that domain.
  The seven component scores are summed to yield a global score ranging from 0 to 21.
  A score of 5 or higher is generally indicative of poor sleep quality.
Evaluate the clinical effect of cannabis extract Avextra 10/10 solution on pain using Widespread pain indexWPI | 4, 8 and 12 weeks
  The WPI lists 19 specific body areas that are grouped anatomically (upper and lower extremities (e.g., shoulders, arms, legs), axial regions (e.g., neck, lower back), cranial and chest regions (e.g., jaw, chest)). These regions are divided into the left and right sides of the body, where applicable.
  The patient indicates whether they have experienced pain in each of these areas during the past week. The response is binary (yes or no) for each area.
  Each body area where pain is reported is assigned a score of 1. The scores from all 19 areas are summed to produce the WPI total score, which ranges from 0 to 19.
Evaluate the effect of cannabis extract Avextra 10/10 solution on the quality of life using The Italian versions of the Revised Fibromyalgia Impact Questionnaire (FIQR) | 4, 8 and 12 weeks
  The Revised Fibromyalgia Impact Questionnaire (FIQR) is a validated, self-administered tool designed to measure the overall impact of fibromyalgia on a patient's daily life. The FIQR consists of 21 questions divided into three main domains:
  * Function (9 items): assesses the patient's ability to perform daily tasks and activities.
  * Overall Impact (2 items): measures the overall effect of fibromyalgia on the patient's life and how they perceive their condition.
  * Symptom Severity (10 items): covers common fibromyalgia symptoms.
  Each question is scored on a 0 to 10 scale, where 0 (No difficulty or symptoms) 10 (Extreme difficulty or worst symptoms).
  The scores from all three domains are combined to give a total FIQR score, ranging from 0 to 100
Describe any adverse events or the principal reasons of drug discontinuation. | 4,8,12 weeks
  Describe any adverse events or the principal reasons of drug discontinuation.
1. Evaluate the clinical effect of cannabis extract Avextra 10/10 solution on pain after 12 weeks among patients affected by FM | 4, 8 weeks
  Description: The secondary endpoint is based on a comparative analysis between the Visual Analogic Scale (VAS) score reported before cannabis extract Avextra 10/10 solution and after 12 weeks of therapy. VAS will use a 100 mm pain line where 0 represents "no pain at all" and 100 is "maximum pain ever experienced".
Evaluate the clinical effect of cannabis extract Avextra 10/10 solution on Functional Appreciation Scale (FAS) | 4, 8, 12 weeks
  The Functional Appreciation Scale (FAS) is a tool designed to assess an individual's overall functionality and their ability to perform daily activities. It evaluates the impact of a condition, such as fibromyalgia, on physical, psychological, and social aspects of functioning. The scale typically captures subjective perceptions of functional limitations, providing valuable insights into the patient's quality of life and the effectiveness of therapeutic interventions
Evaluate the clinical effect of cannabis extract Avextra 10/10 solution on Symptom Severity Scale (SSS) | 4, 8, 12 weeks
  The Symptom Severity Score (SSS) is a tool used to assess the severity of symptoms in conditions like fibromyalgia. It evaluates key symptoms, including fatigue, sleep disturbances, cognitive issues, and somatic complaints, on a scale typically ranging from 0 to 3 (none to severe). The total score reflects the overall symptom burden, helping to classify and monitor the condition's severity.

CONTACTS AND LOCATIONS:
Overall Officials: Piercarlo Sarzi Puttini, Medical Doctor, Principal Investigator — IRCCS Ospedale Galeazzi Sant'Ambrogio
Locations (1):
- IRCCS Ospedale Galeazzi-Sant'Ambrogio, Milan, Milano, Italy

IPD SHARING:
Plan to Share IPD: Yes
The results of this study will be submitted for publication to peer-reviewed journals or for presentation at national and international congresses. Each paper or abstract, must be reviewed and approved by the executive committee prior to submission. IPD will be shared upon reasonable request.

REFERENCES:
- [Background] Sarzi-Puttini P, Giorgi V, Marotto D, Atzeni F. Fibromyalgia: an update on clinical characteristics, aetiopathogenesis and treatment. Nat Rev Rheumatol. 2020 Nov;16(11):645-660. doi: 10.1038/s41584-020-00506-w. Epub 2020 Oct 6. PMID 33024295
- [Background] Pozzi G, Frustaci A, Tedeschi D, Solaroli S, Grandinetti P, Di Nicola M, Janiri L. Coping strategies in a sample of anxiety patients: factorial analysis and associations with psychopathology. Brain Behav. 2015 Aug;5(8):e00351. doi: 10.1002/brb3.351. Epub 2015 Jun 24. PMID 26356192
- [Background] Curcio G, Tempesta D, Scarlata S, Marzano C, Moroni F, Rossini PM, Ferrara M, De Gennaro L. Validity of the Italian version of the Pittsburgh Sleep Quality Index (PSQI). Neurol Sci. 2013 Apr;34(4):511-9. doi: 10.1007/s10072-012-1085-y. Epub 2012 Apr 13. PMID 22526760
- [Background] Cerea S, Todd J, Ghisi M, Mancin P, Swami V. Psychometric properties of an Italian translation of the Functionality Appreciation Scale (FAS). Body Image. 2021 Sep;38:210-218. doi: 10.1016/j.bodyim.2021.04.007. Epub 2021 May 4. PMID 33962221
- [Background] Salaffi F, Franchignoni F, Giordano A, Ciapetti A, Sarzi-Puttini P, Ottonello M. Psychometric characteristics of the Italian version of the revised Fibromyalgia Impact Questionnaire using classical test theory and Rasch analysis. Clin Exp Rheumatol. 2013 Nov-Dec;31(6 Suppl 79):S41-9. Epub 2013 Jun 26. PMID 23806265
- [Background] Sotoodeh R, Waldman LE, Vigano A, Moride Y, Canac-Marquis M, Spilak T, Gamaoun R, Kalaba M, Hachem Y, Beaulieu P, Desroches J, Ware MA, Perez J, Shir Y, Fitzcharles MA, Martel MO. Predictors of Pain Reduction Among Fibromyalgia Patients Using Medical Cannabis: A Long-Term Prospective Cohort Study. Arthritis Care Res (Hoboken). 2023 Jul;75(7):1588-1594. doi: 10.1002/acr.24985. Epub 2023 Feb 3. PMID 35876631
- [Background] Aster HC, Evdokimov D, Braun A, Uceyler N, Sommer C. Analgesic Medication in Fibromyalgia Patients: A Cross-Sectional Study. Pain Res Manag. 2022 Sep 22;2022:1217717. doi: 10.1155/2022/1217717. eCollection 2022. PMID 36247103
- [Background] Chaves C, Bittencourt PCT, Pelegrini A. Ingestion of a THC-Rich Cannabis Oil in People with Fibromyalgia: A Randomized, Double-Blind, Placebo-Controlled Clinical Trial. Pain Med. 2020 Oct 1;21(10):2212-2218. doi: 10.1093/pm/pnaa303. PMID 33118602
- [Background] Giorgi V, Bongiovanni S, Atzeni F, Marotto D, Salaffi F, Sarzi-Puttini P. Adding medical cannabis to standard analgesic treatment for fibromyalgia: a prospective observational study. Clin Exp Rheumatol. 2020 Jan-Feb;38 Suppl 123(1):53-59. Epub 2020 Feb 5. PMID 32116208
- [Background] Mazza M. Medical cannabis for the treatment of fibromyalgia syndrome: a retrospective, open-label case series. J Cannabis Res. 2021 Feb 17;3(1):4. doi: 10.1186/s42238-021-00060-6. PMID 33597032
- [Background] Kurlyandchik I, Tiralongo E, Schloss J. Safety and Efficacy of Medicinal Cannabis in the Treatment of Fibromyalgia: A Systematic Review. J Altern Complement Med. 2021 Mar;27(3):198-213. doi: 10.1089/acm.2020.0331. Epub 2020 Dec 8. PMID 33337931
- [Background] Cameron EC, Hemingway SL. Cannabinoids for fibromyalgia pain: a critical review of recent studies (2015-2019). J Cannabis Res. 2020 May 29;2(1):19. doi: 10.1186/s42238-020-00024-2. PMID 33526114
- [Background] Walitt B, Fitzcharles MA, Hassett AL, Katz RS, Hauser W, Wolfe F. The longitudinal outcome of fibromyalgia: a study of 1555 patients. J Rheumatol. 2011 Oct;38(10):2238-46. doi: 10.3899/jrheum.110026. Epub 2011 Jul 15. PMID 21765102
- [Background] Giorgi V, Sirotti S, Romano ME, Marotto D, Ablin JN, Salaffi F, Sarzi-Puttini P. Fibromyalgia: one year in review 2022. Clin Exp Rheumatol. 2022 Jun;40(6):1065-1072. doi: 10.55563/clinexprheumatol/if9gk2. Epub 2022 Jun 22. PMID 35748720
- [Background] Martinez JE, Guimaraes I. "Fibromyalgia - are there any new approaches?". Best Pract Res Clin Rheumatol. 2024 Mar;38(1):101933. doi: 10.1016/j.berh.2024.101933. Epub 2024 Feb 13. PMID 38355316
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Wolfe F, Smythe HA, Yunus MB, Bennett RM, Bombardier C, Goldenberg DL, Tugwell P, Campbell SM, Abeles M, Clark P, et al. The American College of Rheumatology 1990 Criteria for the Classification of Fibromyalgia. Report of the Multicenter Criteria Committee. Arthritis Rheum. 1990 Feb;33(2):160-72. doi: 10.1002/art.1780330203. PMID 2306288
- [Background] Yellen SB, Cella DF, Webster K, Blendowski C, Kaplan E. Measuring fatigue and other anemia-related symptoms with the Functional Assessment of Cancer Therapy (FACT) measurement system. J Pain Symptom Manage. 1997 Feb;13(2):63-74. doi: 10.1016/s0885-3924(96)00274-6. PMID 9095563
- [Background] Wolfe F, Clauw DJ, Fitzcharles MA, Goldenberg DL, Katz RS, Mease P, Russell AS, Russell IJ, Winfield JB, Yunus MB. The American College of Rheumatology preliminary diagnostic criteria for fibromyalgia and measurement of symptom severity. Arthritis Care Res (Hoboken). 2010 May;62(5):600-10. doi: 10.1002/acr.20140. PMID 20461783